CLINICAL TRIAL: NCT05254028
Title: The Effectiveness of Auricular Point Compared to Body Point Acupuncture Theraphy on Healthcare Workers With Tension-Type Headache in RSUPN Dr. Cipto Mangunkusumo Jakarta
Brief Title: The Effectiveness of Auricular Point Compared to Body Point Acupuncture Theraphy on Tension-Type Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Fieka Meitaqwatiningarum, Principal investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 21-10-1106
Record Dates: First submitted 2022-01-29; First posted 2022-02-24 (Actual); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Tension-Type Headache
Keywords: Acupuncture; Auricular acupuncture; Tension-type headache; Healthcare worker
MeSH Terms: conditions — Tension-Type Headache

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: There will be 4 outcome assessors who do not know the intervention status of study subjects
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular points acupuncture (Active Comparator): The subject of this study is healthcare workers with tension-type headache symptoms who work at Dr. Cipto Mangunkusumo Hospital. The subject of this group will be treated with filiform needles, 30-minute needle retention, 3 times a week for 2 weeks (total of 6 therapy sessions). The "Huanqiu" needles with a size 0.20mm x 13mm are inserted at the auricular acupuncture points shenmen (TF4), thalamus (AT4), and occiput (AT3) bilateral.
  Interventions: Procedure: filiform needle
- Body points acupuncture (Active Comparator): The subject of this study is healthcare workers with tension-type headache symptoms who work at Dr. Cipto Mangunkusumo Hospital. The subject of this group will be treated with filiform needles, 30-minute needle retention, 3 times a week for 2 weeks (total of 6 therapy sessions). The "Huanqiu" needles with a size 0.25mm x 25mm are inserted at the acupuncture points LI4 Hegu, LR3 Taichong, dan GB20 Fengchi bilateral.
  Interventions: Procedure: filiform needle

INTERVENTIONS:
Procedure: filiform needle — Manual acupuncture using filiform needles

SUMMARY:
The purpose of this study is to compare the effectiveness of manual acupuncture between 2 types of points in decreasing tension-type headache symptoms of healthcare workers in Dr.Cipto Mangunkusumo hospital

DETAILED DESCRIPTION:
The purpose of this study is to compare the effectiveness of manual acupuncture therapy between auricular points and body points in improving tension-type headache symptoms based on a headache diary which is consisting of intensity and frequency of headache days, a short form-36 questionnaire, and an examination of the press pressure threshold on eight pericranial muscles. If the use of auricular points is proven to be superior, then this method will benefit the patient more because it is more efficient and can be used as a protocol for providing therapy to patients with tension-type headache.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare workers who work in Dr. Cipto Mangunkusumo hospital
* Age 18-60 years
* Has an episodic or chronic TTH classification and is in accordance with the diagnostic criteria in the International Classification of Headache Disorders 3rd edition beta version (ICHD-3beta)
* Headache with VAS score of 10-70 mm
* Willing to participate in research and sign an informed consent
* Willing to follow the research process to completion.

Exclusion Criteria:

* Migraine headaches or secondary headaches
* Long-term (>10 days per month) uninterrupted use of NSAIDs and other analgesia drugs 24 hours before starting acupuncture therapy
* Has contraindications to acupuncture, namely: medical emergencies, pregnancy, history of bleeding disorders (including the use of anticoagulant drugs) obtained from anamnesis history, tumor, or infection at the acupuncture site.
* Ear deformities and earlobe infections
* Fever 38°C
* Have had acupuncture therapy in the last 7 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2021-12-27 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Headache intensity | 6 weeks
  Headache intensity is recorded in the headache diary, measured by a visual analog score (VAS) consisting of a straight horizontal line numbered 0-100 millimeters (mm) and a description at each end (no pain at 0 mm and very severe pain at 100 mm), then the patient is asked to point a point on the line that corresponds to the degree of pain
Frequency of headache day | 6 weeks
  Frequency of headache day is recorded in the headache diary, as assessed by the presence of headaches > 30 minutes/day.
Pain Pressure Threshold (PPT) | 2 weeks
  PPT is the minimum applied force that can induce pain, in each of 4 bilateral areas: the suboccipital muscle (the insertion of the trapezius muscle), the mid-upper trapezius muscle, the temporal muscle and the splenius capitis muscle. Measurements using the "Weigner" algometer. Measurements in one area were carried out 3 times, with the result being the average of the three.
Short form-36 questionnaire (SF-36) | 6 weeks
  SF-36 is a questionnaire to assess a person's quality of life which consists of 36 questions divided into 8 scales with the results of 2 summary measures, namely physical and mental health. Assessments were carried out using the SF-36 software for scores ranging from 0-100 (0=worst state of health and 100=best state of health). The mean score of 50 was articulated as the normative value for all scales

CONTACTS AND LOCATIONS:
Overall Officials: Fieka Meitaqwatiningarum, dr, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (1):
- Dr. Cipto Mangunkusumo hospital, Jakarta Pusat, DKI Jakarta, Indonesia